CLINICAL TRIAL: NCT06729372
Title: Optimizing Simulation-Based Training in Orthopedics: Exploring Deliberate Flawed Performance for Dynamic Hip Screw Osteosynthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen Academy for Medical Education and Simulation (Other)
Responsible Party: Principal Investigator, Amandus Gustafsson, Associate Professor, Consultant, Ph.D., MD, Copenhagen Academy for Medical Education and Simulation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: F-24069185
Record Dates: First submitted 2024-12-08; First posted 2024-12-11 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Simulation Based Medical Education
Keywords: Deliberate flawed performance; Hip fracture; Simulation-based training
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Error avoidance training (Active Comparator): Participants are instructed to avoid errors during simulation-based training
  Interventions: Behavioral: Error Avoidance Training
- Deliberate flawed training (Active Comparator): The participants are instructed to train deliberate errors during simulation-based training
  Interventions: Behavioral: Deliberate Flawed Performance

INTERVENTIONS:
Behavioral: Deliberate Flawed Performance — Deliberate Flawed Performance during simulation-based training
  Arms: Deliberate flawed training
Behavioral: Error Avoidance Training — Error Avoidance during simulation-based training
  Arms: Error avoidance training

SUMMARY:
Proximal femoral fractures (PFF) are associated with increased mortality when surgical intervention is delayed, with evidence supporting osteosynthesis within 12 to 24 hours of admission to minimize risk.1, 2 Consequently, surgical procedures for PFF should be mastered by orthopedic trainees early in their career. In Denmark, this necessity is reflected in the first-year specialist training curriculum, which designates PFF surgery as one of three procedures requiring mandatory competence assessment.3 From 2013 to 2019, orthopedic trainees performed 66% of all registered PFF surgeries in Denmark.4 However, evidence suggests that surgeries performed by surgeons in training can be associated with higher reoperation rates.2,5,6 Simulation-based training (SBT) has been proposed to reduce this risk, as it is associated with superior learning outcomes compared to other instructional modalities.7 In a Danish national needs assessment of SBT, osteosynthesis for PFF was ranked 2nd of 33 prioritized procedures within orthopedic surgery.8

Simulators for SBT of PFF osteosynthesis are available. One of them is the Swemac TraumaVision simulator and several studies have supplied both supporting validity evidence for the imbedded tests and evidence supported mastery standards for trainees to achieve before continued practice on patients in the operating room under supervision of senior colleagues.9-11 Accordingly, SBT is now part of the Danish national curriculum for specialist training in orthopaedic surgery.12

The training is based on directed self-regulated learning (DSRL), where trainees receive feedback after each iteration of training and use it to improve their performance in subsequent iterations. While DSRL appears to be noninferior to instructor-regulated training,13 experimental studies suggest a potential downside. Feedback given during training may improve immediate performance but can adversely affect long-term retention and the transfer of skills to new settings.14,15 Interestingly, evidence suggests that performing errors during early training may be essential to avoid them in the future16 possibly due to the to the reflection and cognitive activities that errors elicit in the learner.17-19 Further, exploratory behavior during training is shown to have a positive effect on performance outcomes.20 Indeed, evidence from outside the medical field indicates that error management training (EMT), training where errors are pursued and considered desirable for learning, slightly reduces performance during training compared to error avoidance training (EAT) but enhances post training and transfer performance with moderate effect sizes.21-23

Evidence within medical SBT remains limited. However, Dyre et al. have investigated the effect of EMT compared to EAT on medical students' SBT transabdominal fetal ultrasound scans. The students had the same training time, but those who trained with EMT had both statistically and clinically significantly better performance scores and diagnostic abilities on a transfer test on patients, with statistically large and moderate effect sizes, respectively.24 EMT traditionally comprises both an error component and an exploratory component. However, it has been shown that exposure to both correct and flawed performance demonstrations can enhance skill acquisition, provided that learners are informed what errors that the flawed performance contains. The correct example serves as a reference for performance standards, enabling learners to extract meaningful insights from the flawed performance.25,26 A proposed mechanism for this process is that encountering errors compels learners to actively engage with the material, forcing deeper cognitive processing and thereby enhancing training efficacy.27

Hence, there is a sizable knowledge gap as to how EMT may enhance SBT in surgery. It is not clear to what degree the error training component contributes to the perceived positive effects of EMT. Errors made in surgery can be detrimental to patient safety. Accordingly, it is meaningful to explore any method to reduce transfer of such mistakes from training to the clinical setting. Moreover, considering that trainees' time is a valuable and limited resource, and the setup of SBT comes at a cost, it is prudent to explore how these instructional methods may enhance the efficacy of SBT.

The aim of this study is to explore the effect of instructions in deliberate flawed performance (DFP) compared to EAT instructions on retention and transfer of skills on medical students when performing SBT of open surgery in form of osteosynthesis with dynamic hip screw (DHS).

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in medical school at University of Copenhagen passed exam in orthopaedic surgery

Exclusion Criteria:

* prior clinical or simulation-based osteosynthesis experience inability to participate in the transfer and retention test within the designated timeframe after the completion of training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-05-26 (Actual); Study Completion 2025-05-26 (Actual)

PRIMARY OUTCOMES:
Retention test | 7-10 days after training
  Performance on a validated test for the training

SECONDARY OUTCOMES:
Post test | Immediately after training
  Performance on a validated test of the training
Transfer test | 7-10 days after training
  Performance on a validated test for a different, but similar training setup

OTHER OUTCOMES:
Pre-test | Immediately before training
  Performance prior to intervention on a validated test for training

CONTACTS AND LOCATIONS:
Locations (1):
- Copenhagen Academy for Medical Education and Simulation, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided